CLINICAL TRIAL: NCT04968652
Title: Evaluation of the Simplified Diagnosis Tool for Chinese IBS-C (Irritable Bowel Syndrome With Constipation) Patients
Brief Title: IBS-C Questionnaire Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Ruijin Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Henan Provincial People's Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Peking University First Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D5630R00002
Record Dates: First submitted 2021-06-28; First posted 2021-07-20 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Irritable Bowel Syndrome With Constipation; Functional Constipation
Keywords: IBS-C; functional constipation; diagnosis, questionnaire
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS-C Group: Result of ROME VI marked as 'IBS-C'.
- Non IBS-C Group: Result of ROME VI marked as 'Non IBS-C'

SUMMARY:
The study is a multi-centre, observational study which enrolls 150 IBS-C patients and 150 non-IBS-C patients in China.

DETAILED DESCRIPTION:
The potential study subject will be identified by the investigators by face-to-face visit, and there will be only 1 visit in this study. Every patient will complete both ROME IV and the Simplified Diagnosis Tool during the visit, and in the same day.

The study will collect results of the ROME IV and the Simplified Diagnosis Tool. Sensitivity and specificity of simplified diagnosis methodology compared with ROME IV will be analysed after all the data has been collected.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (IBS-C)

* ≥18 years old
* Decrease of frequency of bowel movement (<3 time per week), change of stool consistency (stool that is hard and difficult to pass, Bristol Types 1 to 3), or other 'constipation symptoms' judged by investigators.
* With abdominal symptoms such as abdominal pain, bloating, and abdominal discomfort, or other 'constipation symptoms' judged by investigators.
* Result of ROME VI marked as 'IBS-C'.

Group 2 (non-IBS-C)

* ≥18 years old
* Decrease of frequency of bowel movement (<3 time per week), change of stool consistency (stool that is hard and difficult to pass, Bristol Types 1 to 3), or other 'constipation symptoms' judged by investigators.
* With abdominal symptoms such as abdominal pain, bloating, and abdominal discomfort, or other 'constipation symptoms' judged by investigators.
* Result of ROME VI marked as 'Non IBS-C'.

Exclusion Criteria:

* Individuals with a cognitive condition and unable to finish the questionnaire.
* Individuals have an acute or chronic non-GI condition that can be associated with constipation; e.g., central nervous system cause (Parkinson's disease, spinal cord injury, and multiple sclerosis), pseudo-obstruction, colonic inertia, megacolon, megarectum, bowel obstruction, descending perineum syndrome, solitary rectal ulcer syndrome, systemic sclerosis.
* Individuals who had been diagnosed with the following organic health problems likely to affect GI symptoms:

  * Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
  * cancer anywhere in the GI tract or current infection of the GI tract.
  * Pelvic floor dysfunction. (i.e., disease that is not adequately treated or stable with therapy.)
  * Any history of colon surgeries.
* Individuals who participate in any interventional study currently.
* Not suitable for the study judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: With the ratio of IBS-C/non-IBS-C as 1:1, when the sample size is 300, assuming the sensitivity and specificity using ROME IV as reference are 0.85 and 0.85 respectively, a two-sided 95% confidence interval will produce confidence interval widths of 0.12 and 0.12 respectively.
  In addition, with the same assumption as above, a total sample size of 300 (which includes 150 subjects with the IBS-C) achieves 99% power to detect a change in sensitivity/ specificity from 0.7 to 0.85 using a two-sided binomial test. The target significance level is 0.05.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
the sensitivity and specificity of the Simplified Diagnosis Tool for Chinese IBS-C patients | 14 months
  Sensitivity (%)=(number of patients judged as IBS-C based on both the Simplified Diagnosis Tool and the ROME IV)/( number of patients judged as IBS-C based on ROME IV) ×100% Specificity (%)=(number of patients judged as non-IBS-C based on both the Simplified Diagnosis Tool and ROME IV)/( number of patients judged as non-IBS-C based on The ROME IV) ×100%

SECONDARY OUTCOMES:
the accuracy of the Simplified Diagnosis Tool | 14 month
  Accuracy (%)=(number of patients judged as IBS-C based on both the Simplified Diagnosis Tool and The ROME IV + number of patients judged as non-IBS-C based on both Simplified Diagnosis Tool and The ROME IV) / (total number of patients in the FAS) ×100%
the Kappa coefficient of the Simplified Diagnosis Tool | 14 months
  The Kappa coefficient will be calculated according to the following formula:
  Kappa coefficient=(P0-Pe)/(1-Pe)
the positive predictive value, and negative predictive value of the Simplified Diagnosis Tool | 14 months
  Positive predictive value (%)=(number of patients judged as IBS-C based on both Simplified Diagnosis Tool and The ROME IV)/(number of patients judged as IBS-C based on Simplified Diagnosis Tool) ×100% Negative predictive value (%)=(number of patients judged as non-IBS-C based on both Simplified Diagnosis Tool and The ROME IV)/( number of patients judged as non-IBS-C based on Simplified Diagnosis Tool) ×100%

CONTACTS AND LOCATIONS:
Overall Officials: Lishou Xiong, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (9):
- China (9):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5630R00002&attachmentIdentifier=61fe4bc8-4c5b-4c52-8e85-2a97c863c66e&fileName=Clinical_Study_report_synopsis-IBS-C_-_V1.0_-_20230327.pdf&versionIdentifier=